CLINICAL TRIAL: NCT02246491
Title: Induced Pluripotent Stem (iPS) Cell-Based Approaches For Modeling and Treating Ataxia-Telangiectasia
Brief Title: Cell-Based Approaches For Modeling and Treating Ataxia-Telangiectasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research objectives.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00038916; J1491 (Other: SKCCC)
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Ataxia-Telangiectasia (A-T)
MeSH Terms: conditions — Ataxia Telangiectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPSCs without gene correction (Other): This is not a clinical trial and there is no immediate benefit to the participants. At this time, iPSCs and their derived products are not suitable for administration to patients. However, they are useful for basic and preclinical studies of the disease, such as mechanistic studies of ATM function or screening for small molecules with therapeutic value. As regenerative medicine continues to advance, iPSCs and their products may ultimately be used for clinical studies aimed at replacing damaged tissues in A-T patients.
  Interventions: Other: Carrier patients iPS cell line
- iPSCs with gene correction (Other): This is not a clinical trial and there is no immediate benefit to the participants. At this time, iPSCs and their derived products are not suitable for administration to patients. However, they are useful for basic and preclinical studies of the disease, such as mechanistic studies of ATM function or screening for small molecules with therapeutic value. As regenerative medicine continues to advance, iPSCs and their products may ultimately be used for clinical studies aimed at replacing damaged tissues in A-T patients.
  Interventions: Other: A-T iPS cell line

INTERVENTIONS:
Other: A-T iPS cell line — Reprogramming A-T patients iPS cell line
  Arms: iPSCs with gene correction
Other: Carrier patients iPS cell line — Reprogramming iPS cell line from carrier patients
  Arms: iPSCs without gene correction

SUMMARY:
This research is being done to better understand the causes of the disease Ataxia-Telangiectasia and, in the longer-term, develop new therapies for the disease using stem cells.

Induced pluripotent stem cells (iPSC) are a type of cells that can be made in the laboratory from cells in your body, such as blood cells or skin cells (fibroblasts). These stem cells can then be used for research purposes. For example, stem cells can be used to investigate how the mutation in ATM causes the actual symptoms of Ataxia-Telangiectasia. In addition, the stem cells can be used to screen for drugs that could be helpful to treat the disease or to develop new laboratory techniques to correct the mutation that causes Ataxia-Telangiectasia. where the mutation that causes the disease is corrected by the investigators. The stem cells generated in this study will not be used directly for patient therapy and therefore this research does not have a direct benefit to you. However, it will help advance our understanding of the disease and develop future therapies.

Patients who enroll in this study will get all of the standard therapy they would get for their tumor whether or not they participate in this study. There is no extra or different therapy given. The study involves a one-time procedure (either blood collection or skin biopsy).

DETAILED DESCRIPTION:
Ataxia-Telangiectasia (A-T) is a devastating genetic syndrome of neurodegeneration, immunodeficiency and cancer predisposition caused by mutations in the locus encoding ATM (Ataxia-Telangiectasia Mutated). The current standard of care for A-T consists of aggressive supportive measures, and the prognosis remains poor. There is therefore a pressing need to develop novel experimental approaches and treatments for this disease. In this application, we propose to address this need by developing for the first time human stem cell-based technologies to: 1) generate novel experimental models for A-T that faithfully recapitulate the features of the disease across its complex spectrum of clinical manifestations (Aim 1); and 2) start to test the feasibility of regenerative therapies for A-T, via generation of autologous stem cells that have been rendered disease-free by correction of the mutation (Aim 2). Mutations causing A-T are private, resulting in variable reduction in ATM activity and, correspondingly, a wide spectrum of clinical manifestations. Although the most severe form of the disease ("classical" A-T, with no detectable ATM) has been modeled in the mouse (ATM "knock out"), this approach fails to recapitulate the neurological symptoms of the disease and its characteristic tumor spectrum. Moreover, we are currently lacking experimental models for those patients whose mutations result in reduced ATM activity ("variant" A-T). To address these issues, experiments in Aim 1 will test the hypothesis that the genotype-phenotype correlation in A-T is maintained in patient-derived induced pluripotent stem cells (iPSCs). To test this hypothesis, we will reprogram fibroblasts from A-T patients with variable reduction of ATM levels and determine whether: 1) ATM expression and activity in the iPSCs correlate directly with those observed in the patient fibroblasts they are derived from; 2) the iPSCs recapitulate the phenotypes observed in the fibroblasts, including impaired cell cycle checkpoint activation, defective DNA double-strand break (DSB) repair, radiosensitivity and genomic instability; and 3) these phenotypes in the iPSCs directly correlate with their level of ATM expression/activity. If we find that the genotype-phenotype correlation is maintained in A-T iPSCs, this work would validate a more general use of autologous iPSCs for preclinical studies of A-T, including the evaluation of disease biomarkers, drug testing or genetic screening. The clinical manifestations of A-T result from progressive cell loss and tissue degeneration, making A-T a candidate disease for regenerative therapies. Experiments in Aim 2 will test the hypothesis that correction of the ATM mutation in A-T somatic cells will rescue their severe reprogramming defect and allow the generation of disease-free iPSCs. To test this hypothesis, we propose a series of proof-of-principle experiments using a well-characterized compound heterozygous A-T fibroblast cell line. First, we will "repair" either one or the two ATM mutations in this line by recombination with an exogenous donor plasmid carrying the intact sequence, to generate either "carriers" (one normal allele and one mutated allele) or "intact" cells (two normal alleles). To increase the efficiency of recombination, we will introduce a DSB in close proximity to the mutation using Transcription Activator-Like Effector Nucleases (TALENS) that bind specifically to the mutated region. In Preliminary Experiments, we find that we can successfully induce DSBs and site-specific recombination at a human "safe harbor" locus as well as at the ATM locus itself. After verifying that recombination restores ATM expression and function, we will reprogram the corrected cells into iPSCs and characterize their level of ATM expression, activity and function with passage. Because the "null", "carrier" and "intact" lines are isogenic, the effect of ATM gene dose on reprogramming and iPSC function can be evaluated in these experiments. In this regard, approximately 1% of the US general population is an A-T "carrier", extending the significance of this work well beyond A-T patients. Overall, completion of this Exploratory Project will provide the rationale, expertise and reagents for longer-term studies aimed at modeling and treating A-T with autologous iPSCs and/or their derived products and optimizing the use of regenerative therapies for the general population.

ELIGIBILITY:
Inclusion Criteria:

Patients that meet the classic diagnosis of A-T and for whom the underlying mutation(s) is known. The diagnosis of A-T has been made by the clinician using the following criteria:

1. Characteristic neurological abnormalities, including but not limited to oculomotor apraxia, bulbar dysfunction, postural instability, and ataxia.
2. Presence of telangiectasia on the conjunctivae and/or skin.
3. Laboratory abnormalities including but not limited to elevated serum alpha-feto- protein, level, absence of ATM on western blot, increased x-ray induced chromosomal breakage in comparison to a control population, mutations in both alleles of the ATM gene. Parents of the patients above, who are haploinsufficient and whose mutation is known.

Exclusion Criteria:

Patients under 2 years of age No subjects will be excluded on the basis of age, sex, race, or socio-economic status.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Number of samples of primary A-T fibroblast samples that can be successfully reprogrammed to iPSCs | 2 years
  Fibroblasts from patients with A-T will be collected for eligible, consenting participants and processed for reprogramming and iPSC analysis in the laboratory

SECONDARY OUTCOMES:
Number of samples of patient A-T fibroblasts that can be reprogrammed to iPSCs with and without gene correction | 2 years
  The ATM mutation in patient A-T fibroblasts will be corrected using guided nucleases and the reprogramming efficiency of isogenic corrected and uncorrected fibroblasts will be quantified using standard molecular assays.
Quantification of the cloning efficiency of primary cells haploinsufficient for ATM relative to healthy controls | 2 years
  Fibroblasts from individuals heterozygous for an ATM null mutation will be reprogrammed according to standard protocols and the number of iPSC colonies will be compared to those of healthy controls reprogrammed in parallel.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Franco, M.D., Principal Investigator — SKCCC at Johns Hopkins
Locations (1):
- SKCCC at Johns Hopkins, Baltimore, Maryland, United States